CLINICAL TRIAL: NCT00476970
Title: Improving Colorectal Cancer Screening Rates by Lowering Barriers in Low Income and Non-English Speaking Populations: The Chelsea Colorectal Cancer Screening Project
Brief Title: Colorectal Cancer Screening Navigator Program for Low Income and Non-English Speaking Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sanja Percac-Lima, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2006P 002254
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Cancer Screening; Patient Navigation; Low English Proficiency
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigation Intervention (Experimental): Participants randomized to this arm will receive language-concordant patient navigation in the form of an introductory letter with educational material followed by phone or in-person contact to provide individually tailored interventions.
  Interventions: Behavioral: Patient Navigation
- Usual Care (No Intervention): Participants randomized to this arm will receive no additional navigation beyond the usual care for the duration of the 9-month intervention. Participants will be offered navigation services after the completion of the intervention period.

INTERVENTIONS:
Behavioral: Patient Navigation — Patient navigators will perform an initial interview with participants to identify and explore barriers, work with patients to overcome barriers, educate patients about CRC screening, motivate and coach patients, and schedule and accompany patients to colonoscopy testing
  Arms: Patient Navigation Intervention

SUMMARY:
The goal of this study is to implement and in a controlled randomised trial test a program to identify and overcome barriers to CRC screening and thus improve CRC screening rates at MGH Chelsea HC.

Our hypothesis is that a bilingual navigator program, enhanced by using trained interpreting staff will improve CRC screening rates at MGH Chelsea HC overall, and decrease disparities between patients with limited English proficiency and English speakers

DETAILED DESCRIPTION:
We developed a training program for five health center interpreters fluent in eight different languages. Patients randomly assigned to the study intervention receive an introductory letter in their native language. During the initial contact the navigator educates patients about CRC screening and explores patients' barriers to CRC screening. Based on results from a qualitative study conducted at in 2006, we developed interventions to overcome individual barriers to CRC screening tailored to each individual patient. Specific interventions include elucidation of culturally-specific health beliefs; teaching about cancer risk, colonoscopy, and colon prep administration; and help with appointment-making and transport.

ELIGIBILITY:
Inclusion Criteria:

* Between 52-79 years of age
* Have not had a colonoscopy within the last 10 years
* Have not had a sigmoidoscopy/barium enema within the past 5 years
* Have not had a home fecal occult blood testing within the past year.

Exclusion Criteria:

* Acutely ill
* Dementia
* Metastatic cancer
* Schizophrenia
* Any end stage disease

Ages: 52 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1223 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Eligible Patients In Study and Control Groups Who Undergo CRC Screening | 18 Months

SECONDARY OUTCOMES:
Type of CRC Screening Test Performed in Study vs Control Groups | 18 Months
Number of Polyps and Cancers per 100 Patients in the Study vs Control Group | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Percac-Lima, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Chelsea Health Center, Chelsea, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Percac-Lima S, Grant RW, Green AR, Ashburner JM, Gamba G, Oo S, Richter JM, Atlas SJ. A culturally tailored navigator program for colorectal cancer screening in a community health center: a randomized, controlled trial. J Gen Intern Med. 2009 Feb;24(2):211-7. doi: 10.1007/s11606-008-0864-x. PMID 19067085